CLINICAL TRIAL: NCT02440386
Title: iLink (Incentives for Linkage to ART) Study: A Mixed-methods Study to Improve Linkage to HIV Care
Acronym: iLink
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Cape Town (Other)
Collaborators: Brown University (Other)
Responsible Party: Principal Investigator, Brendan Maughan-Brown, Dr, University of Cape Town
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: HRECREF:849/2014
Record Dates: First submitted 2015-04-24; First posted 2015-05-12 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: HIV

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): The control arm receives standard of care. Standard of care involves referral for ART services and follow-up calls (maximum of 6) to assess whether linkage to care has occurred.
- Incentive (Experimental): The incentive arm receives standard of care plus a R300 voucher. The R300 voucher can be exchanged for cash if the participant starts ART at any clinic of their choice within three months from study enrollment.
  Interventions: Behavioral: Conditional economic incentive

INTERVENTIONS:
Behavioral: Conditional economic incentive — Individuals in the intervention arm will receive the standard of care. In addition, individuals in the intervention arm receive a voucher worth R300. They are told that they will get this money if they:
  1. Initiate ART at any clinic within 3 months from the time of their CD4 count test at the Tutu Tester; and
  2. send a text message to the study team to let us know they have started ART;
  3. Schedule a meeting with a member of the study team to show their clinic card and ARVs to confirm ART initiation.
  Other Names: CEI
  Arms: Incentive

SUMMARY:
The iLink Study examines whether a Conditional Economic Incentive (CEI) may be an effective tool for improving linkage to HIV treatment and care following referral for antiretroviral therapy (ART) services from a mobile health clinic in Cape Town, South Africa. The study examines the feasibility and acceptability of using a R300 (approximately $25 as of April 2015) voucher - that is exchanged for cash upon initiation of ART within 3 months - to increase the uptake of ART among men and women living in low-income areas. This pilot study (n=64) includes a randomised control trial, follow-up telephone calls and medical record reviews, and in-depth interviews.

DETAILED DESCRIPTION:
The initiation of combination antiretroviral therapy (ART) remains a serious challenge globally, and particularly in South Africa, the country with the largest population of people living with HIV worldwide (UNAIDS 2012). South Africa has the largest ART programme globally, yet only half of those needing ART in South Africa were receiving treatment in 2011 (Johnson 2012). Early initiation of ART improves treatment outcomes and reduces AIDS-related morbidity and mortality. Recent studies have demonstrated a secondary benefit of ART in preventing HIV transmission by reducing viral load and thus transmissibility (Cohen et al. 2011; Montaner et al. 2010; Tanser et al. 2013). Despite the personal and public health benefits of ART, South African studies have shown large loss to follow-up at each of the stages required for ART initiation: (1) initial CD4 count testing and returning for results; (2) attending ART readiness counselling; and (3) returning to initiate ART (April et al. 2009; Bassett et al. 2010; Kranzer et al. 2010; Larson et al. 2010; Losina et al. 2010).

Novel interventions are urgently needed to improve linkage to HIV treatment and care post-diagnosis, as increased ART coverage will reduce AIDS-related morbidity and mortality, and HIV incidence. Improving ART coverage is therefore a priority in many regions of the world, and particularly in sub-Saharan Africa, where AIDS remains a key development challenge. Interventions based on theories from the field of behavioural economics, a hybrid of principles from psychology and economics (Bickel et al. 1995), have great potential to help strengthen the contributions of psychology to improving ART outcomes. Conditional economic incentives (CEIs), a financial incentive given upon completion of an outcome that can be objectively measured (i.e. ART initiation), has the potential to leverage two theoretical principles from behavioural economics to improve ART initiation. First, instead of being completely rational and accurate, decision-making is viewed as inherently biased due to a multitude of social-cognitive and affective factors that play a role in cost-benefit analysis, such as emotions, personal beliefs, and contextual factors (Fiske & Taylor 2008). In other words, people's preferred outcomes are largely determined by salient contextual needs (Operario et al. 2013). Second, people have a tendency to give greater value to rewards in the present or near future than those in the more distant future (a phenomenon economists term temporal discounting) and therefore decision-making favours immediate rewards and heavily discounts future outcomes. This poses a challenge for ART initiation as the future benefits of ART may be valued less than an individual's more immediate needs, especially for individuals who currently perceive themselves to be relatively healthy.

A CEI may help overcome this challenge for ART initiation by increasing its immediate benefits. A CEI may therefore help 'nudge' individuals to initiate ART by altering the cost-benefit ratio so that the benefits of ART (i.e. the immediate financial reward and the future health reward) outweigh the immediate costs of ART initiation, such as transport, time off work, long waiting lines and the fear of stigma. The application of CEIs to address HIV prevention and treatment problems is still in its infancy, but they have been successfully employed to improve adherence to ART (Rosen et al. 2007; Sorensen et al. 2007; Javanbakht et al. 2010), increase HIV testing uptake and the collection of HIV tests results (Thornton 2008), and reduce risky sexual behaviours (Baird et al. 2012). This evidence indicates that small incentives-based interventions can 'nudge' individuals towards adopting healthier behaviours.

The proposed research will make a significant contribution to our knowledge about demand creation for HIV treatment and prevention services by examining whether CEIs may also be an effective tool for improving linkage to HIV treatment and care following referral for ART services. The proposed research will examine the feasibility and acceptability of using CEIs to increase the uptake of ART among men and women who are referred for ART services. Our long-term collaborative goal is to utilize the results from this pilot study to prepare a grant application for a fully-powered RCT examining whether CEIs can increase ART initiation.

Objectives To examine the acceptability and feasibility of an incentive intervention aimed at increasing uptake of ART among men and women who are referred for ART (CD4 < 500 or WHO stage 4) by a mobile health clinic.

Acceptability

* Did participants find the randomization process fair and acceptable?
* Was the intervention an incentive that motivated or encouraged uptake of ART?
* Was the incentive amount and type acceptable?
* Were individuals in the control arm discouraged from ART initiation because they felt that their linkage to care efforts were not rewarded?
* Were there cases of patients who were unsatisfied or disappointed as a consequence of the study (eg. they did not receive the incentive, yet they thought they should)?

Feasibility

* Is it possible to recruit men and women into the study on the day of being referred for ART?
* Is it possible to track individuals and recruit individuals for in-depth interviews?
* Is it possible to implement the study as planned:

  * Did the randomization process work?
  * Did participants understand the incentive system?
  * Did participants believe that they would actually receive the incentive?
  * Did the incentive delivery method work?
* What is the potential for individuals to game the incentive system? Did any individuals find a method of receiving the money without starting ART?

Potential Efficacy

* Is ART initiation more likely among men and women who are offered the incentive compared to men and women who are not offered the incentive?
* Is early ART initiation more likely among men and women who are offered the incentive compared to men and women who are not offered the incentive?
* Does retention in care after ART initiation differ among men and women who are offered the incentive compared to men and women not offered the incentive?
* What is the potential for incentives to improve ART initiation given participants behavioural intentions regarding ART initiation and barriers to ART initiation?

ELIGIBILITY:
Inclusion Criteria:

* Referred for ART by the Tutu Tester Mobile Clinic (CD4 ≤ 500 or WHO stage 4)
* Planning to live in the study area for the next 6 months
* Willing and able to provide written informed consent for study participation
* Willing to accept calls from the study staff

Exclusion Criteria:

* Participated in the study previously
* Previously been on ART
* Intoxicated at the time of enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
ART initiation | 3 months
  Commencement of antiretroviral therapy for HIV

SECONDARY OUTCOMES:
Time to ART initiation | 1-52 weeks
  Days between referral for ART and ART initiation
Linkage to Care: first visit to clinic | 3 months
  Self-reported attendance at an HIV/ART clinic within 3 months of study enrollment
Time to linkage to care | 1-52 weeks
  Days between referral for ART and attendance at an HIV/ART clinic
ART retention | 12 months
  Indicator of whether the participant collected his/her ART 1 year after starting treatment
Feasibility - accrual percentage | 6 months
  Number of people enrolled in study/number approached for enrollment
Feasibility - participant tracking | 3 and 6 months post enrolment
  Number of participants contact at 3 and 6 months/number of participants enrolled
Acceptability - adverse events | 6 months
  Unexpected risks/harms of providing incentives as self-reported by participants

CONTACTS AND LOCATIONS:
Overall Officials: Brendan Maughan-Brown, PhD, Principal Investigator — University of Cape Town; Omar Galarraga, PhD, Principal Investigator — Brown University
Locations (1):
- Tutu Tester Mobile Clinic, Desmond Tutu HIV Foundation, Cape Town, Western Cape, South Africa